CLINICAL TRIAL: NCT06471842
Title: Study of the Prevalence of Pediatric Eating Disorders in Inherited Metabolic Diseases With Dietary Treatment
Acronym: MEAL
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240434; 2024-A00172-45 (Other: ID-RCB)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Inherited Metabolism Disease
Keywords: Inherited Metabolism Disease; Paediatric eating disorders; Dietary treatment; Montreal feeding scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Inherited Metabolism Disease (IMD) with dietary treatment: Children with Inherited Metabolism Disease (IMD) with dietary treatment planning to come for a hospital visit (in or out patient) as part of their standard care.
  Interventions: Other: MCH (Montreal Children's Hospital) feeding scale questionnaire and parental questionnaire

INTERVENTIONS:
Other: MCH (Montreal Children's Hospital) feeding scale questionnaire and parental questionnaire — The patient's parents will answer the questionnaire and the investigator will complete the parental questionnaire while asking the questions.

SUMMARY:
The main objective of this study is to estimate the prevalence of Pediatric Eating Disorders (PED) in Inherited Metabolic Diseases (IMD) with dietary treatment between the age of 12 months and 6 years 11 months.

DETAILED DESCRIPTION:
Inherited Metabolic Diseases (IMDs) are rare conditions, which are the consequence of a genetic defect affecting an enzyme or a transporter involved in metabolism. This enzymatic defect leads to the accumulation of a potentially toxic compound located upstream of the deficiency and/or the absence of a compound located downstream of the defect. Treatment is possible and it consists of dietary and/or drug treatment.

Pediatric Eating Disorders (PED) cover "all the difficulties of oral feeding. These may be disorders due to absence of spontaneous feeding behavior, or refusal to eat, and disorders which affect the child's entire psychomotor, language and emotional development.

To date, the investigators note the absence of data on the prevalence of PED in IMDs and more generally on the quality of life and psychomotor development of these patients.

The causes and mechanisms of PED are numerous and heterogeneous. Their origins can be endogenous and/or exogenous.

Our main hypothesis is that the presence of PEDs varies depending on the different categories of IMDs with dietary treatment. Estimating their prevalence would enable awareness and early, better quality care.

This study aims to obtain clear and consistent results from a validated scale. It is a single-site study prospectively including patients from the Necker-Enfants Malades hospital reference center.

Parents will be informed of the study by an investigator (psychomotor therapist or dietician) during a phone call, by email or in hospital prior to the inclusion visit.

On the day of inclusion, the parent's and the child's (depending on their age) non-opposition will be collected before carrying out any procedure and recorded in the patient's medical file.

The MCH (Montreal children's hospital) scale and the parental questionnaire will be proposed by the study investigators at the same time, in a physical interview.

The collection of medical data in the patient's file and the rating of the MCH scale will be done in parallel by the study investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 12 months to 6 years and 11 months old
* Patient with an Inherited Metabolic Diseases with dietary treatment
* Patient having experimented a dietary diversification at least 6 month prior
* Patient whose parents do not object to their participation in the study

Exclusion Criteria:

* Patient with an associated chronic disease
* Patient with diagnosed Autistic Spectrum Disorder (ASD) or Pervasive Developmental Disorders (PDD)
* Patient born before 36 weeks of amenorrhea
* Patient with multiple disabilities
* Patient with dystonia
* Patient with absent or unstable head posture
* Patient whose parents do not fully understand or speak French

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Inherited Metabolism Disease (IMD) with dietary treatment planning to come for a hospital visit as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feeding scale score | 1 day
  MCH (Montreal Children's Hospital) feeding scale score between the age of 12 months and 6 years 11 months.

SECONDARY OUTCOMES:
Disorders severity level differentiation | 1 day
  Differentiation between severe/moderate/mild paediatric eating disorders (PED) using the MCH scale score. This scale makes it possible to differentiate the disorders severity level: mild PED with a score between 61 and 65, moderate PED with a score between 66 and 70 and severe PED with a score higher than or equal to 71.
Paediatric eating disorders prevalence for each pathology | 1 day
  Estimate for each pathology the paediatric eating disorders prevalence using the MCH scale score
Risk factors identification | 1 day
  Identify the paediatric eating disorders' risk factors which are inherent to the disease, environmental and psycho-affective based on the parental questionnaire created for this purpose and the data collected

CONTACTS AND LOCATIONS:
Overall Officials: Manon Tessier, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramsay M, Martel C, Porporino M, Zygmuntowicz C. The Montreal Children's Hospital Feeding Scale: A brief bilingual screening tool for identifying feeding problems. Paediatr Child Health. 2011 Mar;16(3):147-e17. doi: 10.1093/pch/16.3.147. PMID 22379377
- [Background] Evans S, Alroqaiba N, Daly A, Neville C, Davies P, Macdonald A. Feeding difficulties in children with inherited metabolic disorders: a pilot study. J Hum Nutr Diet. 2012 Jun;25(3):209-16. doi: 10.1111/j.1365-277X.2012.01229.x. Epub 2012 Feb 9. PMID 22320889
- [Background] Ouattara A, Resseguier N, Cano A, De Lonlay P, Arnoux JB, Brassier A, Schiff M, Pichard S, Fabre A, Hoebeke C, Guffon N, Fouilhoux A, Broue P, Touati G, Dobbelaere D, Mention K, Labarthe F, Tardieu M, De Parscau L, Feillet F, Bonnemains C, Kuster A, Labrune P, Barth M, Damaj L, Lamireau D, Berbis J, Auquier P, Chabrol B. Individual and Family Determinants for Quality of Life in Parents of Children with Inborn Errors of Metabolism Requiring a Restricted Diet: A Multilevel Analysis Approach. J Pediatr. 2023 Mar;254:39-47.e4. doi: 10.1016/j.jpeds.2022.08.060. Epub 2022 Oct 17. PMID 36265570
- See also: This is the website of the G2M health network, which brings together resources and expertise on hereditary metabolic diseases at national level — https://www.filiere-g2m.fr/
- See also: information website designed by the Oralité group at the Necker-Enfants Malades hospital about paediatric eating disorders — https://www.inforalite.fr/